CLINICAL TRIAL: NCT07132931
Title: Exploring the Efficacy of Mindful Leadership Interventions in Public Administration: A Controlled Trial
Brief Title: Exploring the Efficacy of Mindful Leadership Interventions in Public Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Mª Teresa Navarro Gil, PhD Medicine, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI21/244
Record Dates: First submitted 2025-07-31; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Mindful Leadership

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Leadership Intervention (Experimental)
  Interventions: Behavioral: Mindful Leadership Intervention
- Management Skills Training (Active Comparator)
  Interventions: Behavioral: Management Skills Training

INTERVENTIONS:
Behavioral: Mindful Leadership Intervention — Mindful leadership training program focusing on contemplative practices, mindfulness exercises, and leadership skill development.
  Arms: Mindful Leadership Intervention
Behavioral: Management Skills Training — Standard management skills training including organizational techniques, communication skills, and leadership fundamentals.
  Arms: Management Skills Training

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a mindful leadership intervention compared to a management skills training program in executive staff working in public administration.

The main questions it aims to answer are:

* Does the mindful leadership intervention improve work engagement, transformational leadership, and mental well-being compared to the management skills training?
* What are the effects of these interventions over a six-month follow-up period?

Participants will:

* Be assigned to either a mindful leadership program or a management skills training program.
* Complete assessments measuring leadership qualities, mindfulness, engagement, and well-being before and after the intervention, as well as at six months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Holding managerial positions (Service Chiefs and Section Chiefs from various departments, Groups A1 and A2).
* Length of service in the administration (priority given to longer service).
* Permanent or temporary employment status (priority given to permanent employees).
* Number of training actions undertaken in the last year (priority given to fewer training actions undertaken).

Exclusion Criteria:

* Individuals who requested to participate in the training but did not meet these requirements were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Transformational Leadership (Transformational Leadership Questionnaire) | Baseline (pre-intervention), immediately post-intervention (within 1 week after the last session) and 6-month follow-up.
  Measured using the Spanish adaptation of the Rafferty and Griffin Transformational Leadership Questionnaire (2004; adapted by Salanova et al., 2012). The instrument consists of 15 items grouped into five dimensions (Vision, Inspirational Communication, Intellectual Stimulation, Support, and Recognition), each rated on a 5-point Likert scale from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Total scores range from 15 to 75, with higher scores indicating higher transformational leadership behaviors.

SECONDARY OUTCOMES:
Work Engagement (Utrecht Work Engagement Scale, UWES) | Baseline (pre-intervention), immediately post-intervention (within 1 week after the last session) and 6-month follow-up.
  Measured using the Spanish version of the Utrecht Work Engagement Scale (UWES; Salanova et al., 2001), consisting of 17 items rated from 0 ("Never") to 6 ("Always/Every day"). The scale measures three dimensions: Vigor, Dedication, and Absorption. Total scores range from 0 to 102, with higher scores indicating greater work engagement.
Mindfulness Skills (Five Facet Mindfulness Questionnaire - Short Form, FFMQ-15) | Baseline (pre-intervention), immediately post-intervention (within 1 week after the last session) and 6-month follow-up.
  Measured using the short version of the Five Facet Mindfulness Questionnaire (FFMQ-15; Gu et al., 2016), consisting of 15 items rated on a 5-point Likert scale from 1 ("Never or very rarely true") to 5 ("Very often or always true"). Total scores range from 15 to 75, with higher scores indicating greater mindfulness skills.
Self-Compassion (Self-Compassion Scale - Short Form, SCS-SF) | Baseline (pre-intervention), immediately post-intervention (within 1 week after the last session) and 6-month follow-up.
  Measured using the Spanish version of the Self-Compassion Scale - Short Form (SCS-SF; García-Campayo et al., 2014). The instrument consists of 12 items rated from 1 ("Almost never") to 5 ("Almost always"). Total scores range from 12 to 60, with higher scores indicating greater self-compassion.
Well-being (Pemberton Happiness Index, PHI) | Baseline (pre-intervention), immediately post-intervention (within 1 week after the last session) and 6-month follow-up.
  Measured using the Pemberton Happiness Index (PHI; Hervás & Vázquez, 2013). The first section includes 11 items rated from 0 ("Completely Disagree") to 10 ("Completely Agree"). The second section includes 10 items on daily positive and negative experiences, also rated from 0 to 10. Scores can be combined into a single well-being index ranging from 0 to 10, with higher scores indicating greater well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Finance and Public Administration, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon reasonable request to the corresponding author, subject to approval and data use agreements to ensure participant confidentiality.